CLINICAL TRIAL: NCT07368322
Title: Comparative Analysis of Standard Surgical Techniques vs. "Y Incision" Technique for Aortic Root Enlargement in Patients With Small Aortic Annulus Undergoing Aortic Valve Replacement: A Randomized Open-Label Controlled Trial (CRYSTAL Trial - Comparative Research of Y-Incision vs. Standard Techniques for Aortic Root EnLargement)
Brief Title: Comparative Research of Y-Incision vs. Standard Techniques for Aortic Root EnLargement
Acronym: CRYSTAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: willner nadav MD (Other)
Responsible Party: Sponsor-Investigator, willner nadav MD, Non-Invasive Cardiology Unit Director, Rambam Health Care Campus
Organization: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0337-25-RMB
Record Dates: First submitted 2026-01-08; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Severe Aortic Valve Disease; Aortic Valve Replacement (AVR); Small Aortic Annulus
Keywords: AVR; Aortic Root Enlargement; Small Aortic Annulus; Y Incision
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Intervention Model Description: Y-Incision vs. Standard Techniques for Aortic Root Enlargement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Y-Incision Technique for Aortic Root Enlargement (Experimental): The novel "Y incision" technique by Bo Yang allows implantation of valves up to five sizes larger than the native annulus
  Interventions: Procedure: Y incision Technique (YIT)
- Standard Techniques for Aortic Root Enlargement (Active Comparator): Traditional surgical techniques for aortic root enlargement (ARE), such as the Nicks and Manougian procedures, allow enlargement of only one to two prosthesis sizes and involve complex reconstructive procedures
  Interventions: Procedure: Standard surgical enlargement techniques

INTERVENTIONS:
Procedure: Y incision Technique (YIT) — A "Y"-shaped incision is made from the aortotomy, extending through the left coronary-noncoronary commissure into the aortomitral curtain. Thereafter, a Hemashield patch is sewn to the aortomitral curtain and the undermined aortic annulus, creating a larger space, and the bioprosthetic valve is placed and secured. Finally, the modified aortotomy is closed using the roof technique for better hemostasis and to enlarge the sinotubular junction and proximal ascending aorta. This technique allows the implantation of a valve up to five sizes larger than the native annulus.
  Arms: Y-Incision Technique for Aortic Root Enlargement
Procedure: Standard surgical enlargement techniques — Traditional approaches include aortic root enlargement procedures such as the Nicks, Manougian, and Konno techniques; these procedures aim to widen the annulus and accommodate a larger prosthetic valve, thereby reducing the risk of PPM.
  Arms: Standard Techniques for Aortic Root Enlargement

SUMMARY:
Abstract Background: Aortic valve replacement (AVR) is crucial for patients with severe aortic valve disease. However, managing those with a small aortic annulus (SAA, i.e., annulus diameter < 22 mm) is challenging because implanting a small prosthesis can result in patient-prosthesis mismatch (PPM), suboptimal hemodynamic outcomes, and reduced long-term survival. Traditional surgical techniques for aortic root enlargement (ARE), such as the Nicks and Manougian procedures, have significant limitations, typically allowing enlargement of only one to two prosthesis sizes and involving complex reconstructive procedures. The novel "Y incision" technique by Bo Yang offers a promising alternative, allowing implantation of valves up to five sizes larger than the native annulus, but it lacks comprehensive comparative data on its safety, efficacy, and functional outcomes.

Aim: This study aims to compare the safety outcomes, hemodynamic performance, and functional capacity of the "Y incision" technique versus standard surgical enlargement techniques in patients with a small aortic annulus undergoing AVR, with particular emphasis on objective functional assessment using cardiopulmonary exercise testing (CPET).

Methods: This prospective, randomized, controlled superiority trial will enroll patients with aortic valve disease and a small aortic annulus where conventional AVR is expected to result in moderate or severe PPM. Patients will be randomized 1:1 to either the standard surgical technique group or the "Y incision" technique group. Based on preliminary results and power calculations using the Win Ratio methodology, the sample size is set at 90 patients (45 in each group) to account for potential dropouts.

Primary Endpoint: Hierarchical composite endpoint analyzed using Win Ratio methodology, including (in order of priority): all-cause mortality, stroke, myocardial infarction, total hospitalization rate, moderate or severe PPM, exercise-induced valve dysfunction, and functional improvement at specified time points through 12 months.

Secondary Endpoints: Safety outcomes including intraoperative and 30-day complications, long-term anatomical complications, hemodynamic parameters assessed by echocardiography, functional outcomes measured by 6-minute walk distance and CPET (including peak VO₂), quality of life assessed using KCCQ questionnaire, and prosthetic valve-related outcomes at 3, 6, and 12 months post-surgery.

Conclusion: By providing robust, randomized controlled data with objective functional capacity assessment, this study aims to fill current gaps in knowledge regarding the long-term outcomes, safety profile, and functional benefits of the "Y incision" technique compared to standard surgical methods, potentially establishing evidence-based guidance for managing patients with a small aortic annulus undergoing AVR.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years.
* Patients must have signed and dated an ICF in accordance with regulatory and institutional guidelines before any protocol-related procedures and must be willing and able to comply with scheduled visits.
* Diagnosed with aortic valve disease requiring aortic valve replacement.
* Patients with small aortic annulus relative to body size where conventional AVR result in moderate or severe PPM (defined as cases where the largest prosthesis that can be implanted in the native annulus would provide a predicted iEOA ≤0.85 cm²/m² for BMI <30, or ≤0.70 cm²/m² for BMI ≥30), based on manufacturer specifications and patient BSA).
* Suitable candidates for surgery as determined by the heart team.

Exclusion Criteria:

1. Patients for whom conventional AVR without root enlargement is not expected to result in patient-prosthesis mismatch.
2. Prior cardiac surgery.
3. Severe concomitant valvular disease requiring additional procedures.
4. Active endocarditis.
5. Severe chronic lung disease
6. Pre-existing lower limb deficits or any other medical comorbidities that interfere significantly with gait or the ability to perform exercise testing on a bicycle ergometer
7. Severe left ventricular dysfunction (LVEF < 30%).
8. Contraindications to surgery.
9. Concurrent active treatment in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-04 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite of clinical and functional outcomes (Win Ratio) | At specified time points through 12 months
  A composite hierarchical endpoint analyzed using the Win Ratio methodology. Pairs of patients (one from each study arm) are compared based on a prioritized sequence of outcomes. The hierarchy is: 1. Time to all-cause mortality; 2. Incidence of stroke; 3. Incidence of myocardial infarction; 4. Frequency of total hospitalizations; 5. Presence of moderate/severe Prosthesis-Patient Mismatch (PPM); 6. Exercise-induced valve dysfunction; and 7. Improvement in functional status (defined as ≥1 NYHA class improvement). A "win" is assigned to the patient with the better outcome at each step.
  Win Ratio - The ratio of the total number of wins in the intervention group to the total number of wins in the control group.

SECONDARY OUTCOMES:
Incidence of Major Adverse Events (MAE) through 12 months. | Up to 12 months.
  Number of participants experiencing intraoperative and 30-day complications, and long-term anatomical complications (including valve thrombosis or migration).
  Unit of Measure: Number of participants.
Change in Hemodynamic Parameters (Mean Pressure Gradient). | Baseline, 3, 6, and 12 months.
  Assessment of the prosthetic valve mean pressure gradient as measured by transthoracic echocardiography.
  Unit of Measure: mmHg.
Change in 6-Minute Walk Distance (6MWD). | Baseline and 12 months.
  Change from baseline in the distance walked during a 6-minute period. Unit of Measure: Meters.
Change in Quality of Life (KCCQ-12 Score). | Baseline, 3, 6, and 12 months.
  Change in the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) overall summary score. Scores range from 0 to 100, where higher scores represent better health status.
  Unit of Measure: Points on a scale.
Change in Peak Oxygen Consumption (Peak VO2) | Baseline and 12 months post-surgery.
  Peak VO2 attained during Cardiopulmonary Exercise Testing (CPET) using a standardized ramp protocol on a cycle ergometer or treadmill. Unit of Measure: mL/kg/min
Incidence of Prosthetic Valve-Related Complications | 3, 6, and 12 months post-surgery.
  Number of participants experiencing specific valve-related adverse events, including prosthetic valve thrombosis, device migration, endocarditis, or structural valve deterioration (SVD) as defined by VARC-3 criteria.
  Unit of Measure: Number of participants
Incidence of Early Postoperative Complications (30 Days) | Within 30 days post-surgery.
  A composite of safety events occurring within the early postoperative period, including major bleeding (BARC type 3 or 5), acute kidney injury (Stage 2 or 3), and new-onset permanent atrial fibrillation.
  Unit of Measure: Number of participants
Change in Effective Orifice Area (EOA) | Baseline, 3, 6, and 12 months post-surgery.
  The Effective Orifice Area of the prosthetic valve calculated via the continuity equation using transthoracic echocardiography (TTE) measurements. Unit of Measure: cm^2
Change in NYHA Functional Classification | Baseline, 3, 6, and 12 months post-surgery.
  Assessment of heart failure symptoms according to the New York Heart Association (NYHA) Functional Classification. Scores range from Class I (no symptoms) to Class IV (severe symptoms).
  Unit of Measure: NYHA Class (I, II, III, or IV)

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Undecided